CLINICAL TRIAL: NCT01273948
Title: A Randomized, Active-Control Phase II Pilot Trial of Bavituximab Combined With Ribavirin for Initial Treatment of Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Pilot Trial of Bavituximab Combined With Ribavirin for Initial Treatment of Chronic HepC Virus Genotype 1 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 1003
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — bavituximab; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bavituximab 3 mg/kg (Experimental): Bavituximab 3 mg/kg given by intravenous (IV) infusion once weekly, plus oral ribavirin 1000 mg (weight <75 kg) or 1200 mg (weight greater than or equal to 75 kg) divided into twice-daily doses, for 12 weeks
  Interventions: Drug: Bavituximab
- Bavituximab 0.3 mg/kg (Experimental): Bavituximab 0.3 mg/kg given by IV infusion once weekly, plus oral ribavirin 1000 mg (weight <75 kg) or 1200 mg (weight greater than or equal to 75 kg) divided into twice-daily doses, for 12 weeks
  Interventions: Drug: Bavituximab
- Pegylated interferon (PEG-IFN) (Active Comparator): Pegylated interferon (PEG-IFN) alpha-2a 180 micrograms given by subcutaneous (SC) injection once weekly, plus oral ribavirin 1000 mg (weight <75 kg) or 1200 mg (weight greater than or equal to 75 kg) divided into twice-daily doses, for 12 weeks
  Interventions: Drug: Pegylated interferon (PEG-IFN)

INTERVENTIONS:
Drug: Bavituximab — 1. Bavituximab 3 mg/kg given by intravenous (IV) infusion once weekly, plus oral ribavirin 1000 mg (weight <75 kg) or 1200 mg (weight greater than or equal to 75 kg) divided into twice-daily doses, for 12 weeks or
  2. Bavituximab 0.3 mg/kg given by IV infusion once weekly, plus oral ribavirin 1000 mg (weight <75 kg) or 1200 mg (weight greater than or equal to 75 kg) divided into twice-daily doses, for 12 weeks or
  Other Names: Bavituxmab
  Arms: Bavituximab 0.3 mg/kg; Bavituximab 3 mg/kg
Drug: Pegylated interferon (PEG-IFN) — Pegylated interferon (PEG-IFN) alpha-2a 180 micrograms given by subcutaneous (SC) injection once weekly, plus oral ribavirin 1000 mg (weight <75 kg) or 1200 mg (weight greater than or equal 75 kg) divided into twice-daily doses, for 12 weeks
  Other Names: Pegasys
  Arms: Pegylated interferon (PEG-IFN)

SUMMARY:
This will be a randomized, open-label, active-control Phase II pilot trial of bavituximab combined with ribavirin for initial treatment of chronic HCV genotype 1 infection. Eligible patients with normal coagulation, hematological, and renal function will undergo a screening/washout period of up to 28 days, followed by randomization to receive weekly bavituximab or PEG-IFN alpha-2a therapy for 12 weeks, both with twice-daily ribavirin.

The primary endpoint of this study is the proportion of patients who show a greater than or equal to 2-log10 IU reduction in plasma HCV RNA level after 12 weeks of treatment (early virological response; EVR).

Secondary endpoints include the proportion of patients with an undetectable HCV RNA level after 12 weeks of treatment; the proportion of patients who show a reduction in HCV RNA level of greater than or equal to 2 log10 IU after 4 weeks of treatment, viral kinetics for individual patients over time, and comprehensive evaluation of the safety and tolerability of bavituximab infusion.

DETAILED DESCRIPTION:
Primary Objective: The primary objective of this study is to assess the effect of 12 weeks of initial treatment with bavituximab versus PEG-IFN, each combined with ribavirin, on plasma HCV RNA level in patients with chronic HCV genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 65 years
2. Chronic hepatitis C virus (HCV) genotype 1 infection
3. HCV RNA level >10,000 IU/mL
4. Chronic HCV infection, defined as:

   * Previous documentation of positive HCV serology (HCV antibody or RNA) at least 6 months (24 weeks) previously, or
   * Positive HCV serology (HCV antibody or RNA) with a prior remote (more than 6 months previously) risk factor for acquisition of HCV or
   * Historical biopsy consistent with chronic HCV infection
5. No clinically significant abnormalities in hematology, coagulation, or chemistry variables:

   * Hemoglobin >12 g/dL for women; >13 g/dL for men
   * Total white cell count >3000/mm3 and absolute neutrophil count >1500/mm3
   * Platelets >100,000/mm3
   * Prothrombin time (PT) and/or international normalized ratio (INR) less than or equal to 1.2 times the local upper limit of normal (ULN)
   * Conjugated (direct) bilirubin less than or equal to 1.5 times the ULN
   * Serum creatinine within normal limits
   * Thyroid-stimulating hormone (TSH) and free thyroxine (T4) within normal limits
6. Female patients: negative urine pregnancy test
7. Ability to provide informed consent

Exclusion Criteria:

1. Previous interferon-based antiviral therapy for chronic HCV infection
2. Previous treatment with known immunogenic drugs
3. Concomitant human immunodeficiency (HIV) or hepatitis B virus (HBV) infection
4. Cause of liver disease other than chronic HCV infection, such as autoimmune or alcoholic liver disease
5. Decompensated clinical liver disease, including a history of encephalopathy, bleeding esophageal or gastric varices, or ascites
6. Recipient of liver or other solid-organ transplantation
7. Evidence of clinically significant bleeding, defined as gross hematuria, hemoptysis, or gastrointestinal bleeding
8. History of bleeding diathesis or coagulopathy (eg, von Willebrand disease or hemophilia)
9. History of thromboembolic events (eg, deep-vein thrombosis [DVT] or pulmonary embolism). Previous central venous catheter-related thrombosis is acceptable if there is resolution recorded at least 12 months before enrollment.
10. Requirement for concurrent treatment with oral or parenteral anticoagulants or hormones (estrogen-containing contraceptives, hormone replacement, antiestrogen agents, progestins)
11. Condition requiring daily therapy with antiplatelet agents (eg, thienopyridines, dipyridamole, cilostazol; cardiovascular prophylaxis with aspirin is allowed) or corticosteroids
12. Investigational therapy within 28 days before the first planned dose of study drug
13. Major surgery within 28 days before the first planned dose of study drug
14. Uncontrolled intercurrent disease (eg, diabetes, hypertension, thyroid disease)
15. Ongoing angina pectoris or other symptoms of coronary artery disease (CAD); history of stroke, or transient ischemic attack (TIA)
16. History of suicidal ideation or attempt
17. Condition requiring treatment (past or current) with coumarin-type agents
18. Cardiac arrhythmia requiring medical therapy
19. Serious nonhealing wound (including wound healing by secondary intention, ulcer, or bone fracture)
20. Cancer, autoimmune disease, or any disease or concurrent therapy known to cause significant alteration in immune function (corticosteroids are allowed before study enrollment and during the study to treat an AE)
21. Female patients and female partners of male patients: pregnancy, lactation, or inability/unwillingness to practice effective contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in Hepatitis C Virus RNA | 12 weeks
  The primary endpoint is the proportion of patients who show a greater or equal 2-log(10) IU reduction in HCV RNA level at Study Week 12 (early virological response, EVR).

CONTACTS AND LOCATIONS:
Overall Officials: Janet Nuttall, MPH, Study Chair — Peregrine Pharmaceuticals
Locations (1):
- LTD Vakhtang Bochorishvili Anticeptic Centre, Tbilisi, Georgia